CLINICAL TRIAL: NCT03241615
Title: The Relationship Between Dysphagia Symptom Severity and Quality of Life
Brief Title: Dysphagia Symptom Severity and Quality of Life
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Other Study IDs: HACETTEPEUNIVERSITY
Record Dates: First submitted 2017-08-03; First posted 2017-08-07 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Neurogenic Dysphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurogenic dysphagia: Patients with neurogenic dysphagia who will willing to participate in the study, being over the age of 18, normal cognitive function ([24 points according to the Mini Mental State Examination), suffering from dysphagia at least one month, and having clinically stable neurological disease will be included. Dysphagia evaluation will be performed.
  Interventions: Other: Dysphagia evaluation

INTERVENTIONS:
Other: Dysphagia evaluation — Dysphagia evaluation is performed in a clinical setting by an eating assessment tool. Swallowing related quality of life is also assessed.

SUMMARY:
The aim of the study is to investigate the relationship between dysphagia symptom severity and quality of life of the patients with neurogenic dysphagia.

DETAILED DESCRIPTION:
The dysphagia related quality of life and perceived dysphagia symptom severity by patients will be used as a complementary information on oropharyngeal dysphagia. Thus, the aim of the study is to investigate the relationship between dysphagia symptom severity and quality of life of the patients with neurogenic dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study
* Being over the age of 20
* Normal cognitive function
* Suffering from dysphagia at least one month

Exclusion Criteria:

* Being under the age of 20 and above 65 years.
* Abnormal cognitive function
* Clinically unstable neurological disease

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have neurogenic dysphagia and willing to participate in the study, being over the age of 20, normal cognitive function (24 points according to the Mini Mental State Examination), and having clinically stable neurological disease will be included.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Dysphagia symptom severity | 1 month
  Dysphagia symptom severity will be determined by an eating assessment tool.

SECONDARY OUTCOMES:
Quality of life assessment | 1 month
  Swallowing related quality of life will be determined by an dysphagia specific quality of life instrument called Swallow Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No